CLINICAL TRIAL: NCT07078071
Title: Clinical Trial for Evaluating the Effectiveness and Safety of the Pulse Wave-based Atrial Fibrillation and Premature Beat Alert Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huawei Device Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HW-XLSCRJ-001
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Arrhythmia, Heart
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Electrocardiography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atrial Fibrillation (Experimental)
  Interventions: Device: ECG
- Premature beats (Experimental)
  Interventions: Device: ECG
- No evidence of atrial fibrillation/premature beats (Experimental)
  Interventions: Device: ECG

INTERVENTIONS:
Device: ECG — Each participant undergoes testing with both the investigation device and the control device simultaneously. The results of the investigation device, which are obtained through pulse wave data analysis at the wrist, are compared to the investigator's interpretation of the ECG.

SUMMARY:
This study aims to validate the efficacy and safety of the Pulse Wave-based Atrial Fibrillation and Premature Beat Alert Software (Huawei Device Co., Ltd.). This software can provide alerts, store and display PPG data transmitted from smartwatches or fitness trackers. The software is limited to alerting of atrial fibrillation and premature beat, and the results are only for clinical reference.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old, regardless of gender;
2. Participants who meet one of the following conditions according to the medical history in the past 3 months or the ECG during the screening period:

   1. Patients with normal sinus rhythm;
   2. Patients with persistent or permanent paroxysmal atrial fibrillation or in the onset of paroxysmal atrial fibrillation;
   3. Patients with frequent premature beats (more than 5 per minute) or in the onset of premature beats;
3. Patients who volunteer to participate and have signed an informed consent form.

Exclusion Criteria:

1. Patients using cardiac pacemakers or implantable cardioverter defibrillators (ICD);
2. Patients with non-respiratory sinus arrhythmia, sinus arrest or sick sinus syndrome according to the ECG results during the screening period;
3. Patients with interpolated premature beats, junctional premature beats, or escape rhythms according to the ECG results during the screening period;
4. Patients with atrial flutter, ventricular flutter, or ventricular fibrillation according to the ECG results during the screening period;
5. Patients with atrial fibrillation or premature beats who have a resting heart rate of slower than 50 beats/minute or faster than 110 beats/minute according to the ECG results during the screening period;
6. Patients who are critically ill, making it difficult to make an accurate assessment of the effectiveness and safety of the device;
7. Patients who suffer from tremor diseases or chorea, making it difficult to complete the examination quietly;
8. Patients with bullous diseases or large-area skin rashes that are not suitable for body surface electrode recording;
9. Patients whose skin is allergic to ethanol;
10. Patients with contagious skin diseases;
11. Patients with tattoos on their wrist skin that is to be measured;
12. Patients with poor compliance who are unable to cooperate to complete this investigation on their own;
13. Patients who have participated in other clinical investigations within the past 30 days that may affect this investigation;
14. Other conditions that the investigators consider inappropriate for participation in the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of atrial fibrillation identification in a single measurement | 45seconds
Sensitivity and specificity of premature beat identification in a single measurement | 45seconds

SECONDARY OUTCOMES:
Accuracy in identifying the non-arrhythmia in a single measurement | 45seconds
Total identification compliance rate in a single measurement | 45seconds
Software usability | 45seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, China